CLINICAL TRIAL: NCT06828692
Title: Implementation of Machine Learning and Hemodynamic Profiles Based Clinical Decision Support Systems for Personalized Guideline Accordant Antihypertensive Regimens in Primary Care: a Pragmatic Cluster Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCRCSZ-2023-014
Record Dates: First submitted 2025-02-06; First posted 2025-02-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypertension
Keywords: Hypertension; CDSS; cluster randomized controlled trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (CG+ML) (Experimental)
  Interventions: Combination Product: Group A (clinical guideline+machine learning)
- Group B (CG+ICG+ML) (Experimental)
  Interventions: Combination Product: Group B (clinical guideline+impedance cardiograph+machine learning)
- Group C (UC) (Other)
  Interventions: Other: Group C (usual care)

INTERVENTIONS:
Combination Product: Group A (clinical guideline+machine learning) — Group A (CG+ML): A Clinical Decision Support System (CDSS) with the algorithm that incorporates clinical guideline (CG) and machine learning (ML) approach.
  Arms: Group A (CG+ML)
Combination Product: Group B (clinical guideline+impedance cardiograph+machine learning) — Group B (CG+ICG+ML): A Clinical Decision Support System (CDSS) with the algorithm that incorporates clinical guideline (CG), hemodynamic parameters measured by impedance cardiograph (ICG), and machine learning (ML) approach.
  Arms: Group B (CG+ICG+ML)
Other: Group C (usual care) — Control group, the physicians manage the hypertensive patients according to their knowledge and experiences.
  Arms: Group C (UC)

SUMMARY:
This trial is a prospective, multicenter, single-blind, three-arm parallel-group, cluster randomized controlled trial assessing the effectiveness and safety of two types of CDSS in primary care settings in China. Primary care sites are randomized to one of the intervention arms or the control arm (1:1:1 ratio) using computer-generated random numbers stratified by region and administrative categories of the primary healthcare institutions (including community health centers, community health stations, and township health centers). A total of 51 primary care sites are randomized to three groups, with 17 sites assigned to group A (use a CDSS based on clinical guidelines and machine learning), 17 sites to group B (use a CDSS based on guidelines, hemodynamic parameters and ML), and the remaining 17 sites to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. 35 ≤ Age < 80 years.
2. Regularly attend the clinic for hypertension treatment during the study period, without plans of traveling during the study period.
3. Diagnosed with hypertension, with SBP ≥140mmHg at screening.
4. Currently taking 0 or 2 classes of antihypertensive medications (A/C/D), with or without concurrent use of class B.
5. Willing to participate in the trial and capable of providing written informed consent.

Exclusion Criteria:

1. Physician-diagnosed or suspected secondary hypertension (e.g., hypertension caused by renal disease, renal artery stenosis, aortic stenosis, primary aldosteronism, pheochromocytoma/paraganglioma, Cushing's syndrome, thyroid dysfunction, intracranial disease, drug-induced, or rare monogenic genetic disease).
2. SBP ≥180mmHg and/or DBP ≥110mmHg at the screening visit.
3. Suspected or diagnosed white coat hypertension.
4. History of coronary heart disease.
5. History of heart failure.
6. Intolerance to 2 or more classes of A, C,D antihypertensive medications.
7. Currently taking antihypertensive medications other than class A,B,C and D.
8. Diagnosed chronic kidney disease, estimating Glomerular Filtration Rate (eGFR)< 60 ml/min·1.73m2, or receiving dialysis.
9. Serious medical conditions (e.g., malignant cancer and hepatic dysfunction)
10. Currently in an acute episode of disease (e.g, new-onset cardiovascular and cerebrovascular disease occurred within 3 months).
11. Cognitive or communicative disorders.
12. Currently pregnant or breastfeeding or planning a pregnant or breastfeeding during the study.
13. Reluctant to take antihypertensive medications or have poor compliance with previous treatment.
14. Participating in other clinical trials.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
hierarchical composite outcome | Baseline; 3 months
  The primary outcome of the trial is a hierarchical composite outcome, evaluated using the Win-ratio method in the following order:
  1. Office blood pressure control rate (<130/80 mmHg) at 3 months after randomization.
  2. The duration from baseline to the first occurrence of controlled blood pressure achievement (<130/80 mmHg) within 3 months after randomization.
  3. The composite index of the number and dosage of antihypertensive drugs among participants achieved controlled blood pressure at 3 months after randomization.

SECONDARY OUTCOMES:
Separate evaluation of each component of the three-tier hierarchical composite primary outcome at 3 months | Baseline; 3 months
Changes in office systolic and diastolic blood pressure from baseline to 1 month and 3 months | Baseline; 1 month; 3 months
Average 24-hour ambulatory systolic and diastolic blood pressure, along with blood pressure control rate at 3 months | 3 months
Changes in hemodynamic parameters measured by ICG from baseline to 3 months | Baseline; 3 months
  Including dynamic parameters (heart rate and cardiac index), resistance parameters (arterial stiffness index and systemic vascular resistance index), and volume parameters (thoracic blood volume saturation)
Differences in the three-tier hierarchical composite primary outcomes and each component of the three-tier hierarchical composite primary outcome among intervention groups at 3 months | Baseline; 3 months

OTHER OUTCOMES:
safety outcome | Baseline; 3 months
  Safety outcomes include serious adverse events, non-serious adverse events, such as symptomatic hypotension or SBP <90 mmHg, injury falls, syncope, and bradycardia (heart rate <50 beats/minute) during study periods.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zheng, Principal Investigator — Fuwai Hospital, China Academy of Medical Sciences, National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Shenzhen Hospital, Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, China